CLINICAL TRIAL: NCT04271735
Title: Pilot Study to Evaluate the Effect of Nicotinamide Riboside on Immune Activation in Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 200044; 20-H-0044
Record Dates: First submitted 2020-02-14; First posted 2020-02-17 (Actual); Results first posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-03

CONDITIONS: Psoriasis; Atherosclerotic Cardiovascular Disease; Obesity; Dyslipidemia; Cardiometabolic Diseases
Keywords: Chronic Inflammatory Skin Disease; Systemic Inflammation-Induced Atherosclerosis; TH17 Cell Cytokine IL-17 Secretion in Response to T-cell Differentiation; Effect of NR on Neutrophils; Effect of NR on HDL
MeSH Terms: conditions — Psoriasis; Atherosclerosis; Obesity; Dyslipidemias | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants with mild to moderate Psoriasis receiving Placebo (Placebo Comparator): Participants with mild to moderate Psoriasis receiving placebo (2 capsules) twice daily by mouth for 28 days.
  Interventions: Other: Placebo
- Participants with mild to moderate Psoriasis receiving Nicotinamide Riboside (Experimental): Participants with mild to moderate Psoriasis receiving Nicotinamide Riboside Chloride 500mg (2 capsules) twice daily by mouth for 28 days.
  Interventions: Dietary Supplement: Niagen

INTERVENTIONS:
Dietary Supplement: Niagen — Participants will take two capsules of nicotinamide riboside (NR) by mouth (250mg NR or placebo) twice daily for a total of 4 weeks.
  Other Names: Nicotinamide Riboside Chloride; Nicotinamide Riboside
  Arms: Participants with mild to moderate Psoriasis receiving Nicotinamide Riboside
Other: Placebo — Placebo capsule to match the active supplement. Participants will take two capsules, twice daily for a total of 4 weeks.
  Arms: Participants with mild to moderate Psoriasis receiving Placebo

SUMMARY:
Background:

Psoriasis causes chronic inflammation in the body. Researchers want to see if a kind of vitamin B3 dietary supplement can help. This might lead to more treatment options.

Objective:

To test if the dietary supplement nicotinamide riboside can improve immune system function in the blood and skin of people with mild to moderate psoriasis.

Eligibility:

People ages 18-80 with mild to moderate active psoriasis not currently treated with biological therapy

Design:

Participations will be screened with:

* Medical and medication history
* Physical exam
* Measure of body mass index
* Skin exam
* Blood and urine tests

Participants will have visit 1. They will have repeats of the screening tests. They may also have 2 skin biopsies, which are optional. These will be from both lesions and unaffected areas. The areas will be injected with a numbing medicine. A round cutting device will remove small pieces of skin from each area.

Participants will take the study supplement or a placebo starting at the first visit. Neither participants nor the study team will know which they receive. Participants will take capsules twice daily for a total of 4 weeks.

Participants will then have visit 2. This will include the tests performed at visit 1.

Participants may by contacted by phone or email between visits to see how they are doing.

If participants develop any side effects in the 7 days after they stop taking the capsules, they may have another visit.

DETAILED DESCRIPTION:
Study Description:

Psoriasis is a Th17 linked inflammatory disease and we find that the vitamin B3 analogue nicotinamide riboside (NR) blunts Th1 and Th17 activation in ex-vivo na(SqrRoot) ve and differentiated T cells from control and psoriasis subjects. These findings supported the proposal of the following hypothesis. Supplementation with NR will blunt systemic immune activation in mild/moderate psoriasis.

Objectives:

1) Evaluate the effect of NR on Th17 biology

Endpoints:

The primary outcome will be the change in the TH17 cell cytokine IL-17 secretion in response to T-cell differentiation comparing the baseline versus NR or placebo. The comparisons will be performed using paired two-tailed Student t-tests. Significance will be tested at the 0.05 alpha level in this pilot study.

Exploratory outcomes are:

1. Evaluate the effect of NR on the T cell transcriptome
2. Explore the effect of NR on low-density granulocytes and neutrophils

Study Population:

Up to 40 male and female subjects of all races between the ages of 18-80 years with mild-moderate psoriasis who live locally will be screened.

Enrollment and study visits will take place at the NIH Clinical Center or via telehealth visits.

Enrolling Participants:

Psoriatic Subjects

Description of Study Intervention:

Nicotinamide Riboside Chloride 500mg or placebo twice daily by mouth for 28 days.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals must meet all inclusion criteria listed below in order to be eligible to participate in the study.

* Males and females between the ages of 18 and 80 with mild to moderate active psoriasis.
* Female subjects of child-bearing ability willing to commit to reliable contraception while participating in the study.
* Ability to provide informed consent
* Willingness and ability to participate in required study procedures

EXCLUSION CRITERIA:

* Severe psoriasis by PASI (Psoriasis Area and Severity Index) score > 12
* Currently being treated with biologic immune modifying agents.
* Currently on treatment for allergies or other inflammatory diseases.
* Currently taking a multivitamin, Vitamin B or tryptophan supplementation and unwilling to stop within 2 weeks of baseline visit.
* Unwillingness/inability to provide informed consent
* ALT > x3 upper limit of normal, hepatic insufficiency or active liver disease
* Recent history of acute gout
* Chronic renal insufficiency with creatinine > 2.5mg/dl
* Pregnant (or attempting to become pregnant) women
* Current participation in another drug study
* History of intolerance to NR precursor compounds, including niacin or nicotinamide
* Study adherence concerns
* Individuals with diabetes type 1 and 2 who use insulin
* Women of child-bearing potential unwilling to use contraception or unwilling to practice abstinence
* Breastfeeding women unwilling to stop breastfeeding
* Immunization administered within 30 days of participation and no plans for immunization while participating in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael N Sack, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-H-0044.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants With Mild to Moderate Psoriasis Receiving Nicotinamide Riboside | Participants With Mild to Moderate Psoriasis Receiving Placebo
Started | 17 | 12
Completed | 15 | 12
Not Completed | 2 | 0
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Mild to Moderate Psoriasis Receiving Nicotinamide Riboside | Participants With Mild to Moderate Psoriasis Receiving Placebo | Total
Number analyzed (Participants) | 17 | 12 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 10 | 24
  >=65 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 12 | 6 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 15 | 8 | 23
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 13 | 9 | 22
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 17 | 12 | 29

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in the TH17 Cell Cytokine IL-17 Secretion in Response to T-cell Differentiation
Description: Mean change in the TH17 cell cytokine IL-17 secretion in response to T-cell differentiation comparing the baseline versus NR or placebo.
Time Frame: Baseline and Day 28
Population: One participant from placebo group not included in analysis due to insufficient T-cells. One participant from Nicotinamide Riboside group not included in analysis due to abnormal lipids.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Participants With Mild to Moderate Psoriasis Receiving Nicotinamide Riboside | Participants With Mild to Moderate Psoriasis Receiving Placebo
Number analyzed (Participants) | 14 | 11
pg/mL | -176.9 (174.7) | -7.2 (120.9)
Statistical Analysis 1: Comparison: Participants With Mild to Moderate Psoriasis Receiving Nicotinamide Riboside vs Participants With Mild to Moderate Psoriasis Receiving Placebo; Test type: Superiority; p = 0.01, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to day 35
Description: Grade 2 - 5 adverse events and serious adverse events whether volunteered by the patient, discovered by study personnel during questioning, or detected through physical examination, clinically significant laboratory test, or other means will be recorded.
Arm/Group | Participants With Mild to Moderate Psoriasis Receiving Nicotinamide Riboside | Participants With Mild to Moderate Psoriasis Receiving Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/12
Other Adverse Events (participants affected / at risk) | 1/17 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Mild to Moderate Psoriasis Receiving Nicotinamide Riboside (N=17) | Participants With Mild to Moderate Psoriasis Receiving Placebo (N=12)
Fatigue (General disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/35/NCT04271735/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-16): https://cdn.clinicaltrials.gov/large-docs/35/NCT04271735/ICF_001.pdf